CLINICAL TRIAL: NCT04005716
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study of Platinum Plus Etoposide With or Without Tislelizumab (BGB-A317) in Patients With Untreated Extensive-Stage Small Cell Lung Cancer
Brief Title: Study of Platinum Plus Etoposide With or Without Tislelizumab in Participants With Untreated Extensive-Stage Small Cell Lung Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BGB-A317-312; CTR20190511 (Registry Identifier: ChinaDrugTrials)
Record Dates: First submitted 2019-07-01; First posted 2019-07-02 (Actual); Results first posted 2025-02-28 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — tislelizumab; Cisplatin; Carboplatin; Etoposide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A: Tislelizumab + Chemotherapy (Experimental): Participants received tislelizumab in combination with either cisplatin or carboplatin (at the investigator's discretion) and etoposide during the induction phase, administered every 3 weeks for 4 cycles. Upon completion of the induction phase, participants transitioned to maintenance therapy with tislelizumab only, administered once every 3 weeks.
  Interventions: Drug: Tislelizumab; Drug: Cisplatin; Drug: Carboplatin; Drug: Etoposide
- Arm B: Placebo + Chemotherapy (Placebo Comparator): Participants received a placebo in combination with either cisplatin or carboplatin (at the investigator's discretion) and etoposide during the induction phase, given every 3 weeks for 4 cycles. Upon completion of the induction phase, participants transitioned to maintenance therapy with placebo only, administered once every 3 weeks.
  Interventions: Drug: Cisplatin; Drug: Carboplatin; Drug: Etoposide; Drug: Placebo

INTERVENTIONS:
Drug: Tislelizumab — 200 mg administered intravenously on Day 1 of each 21-day cycle
  Arms: Arm A: Tislelizumab + Chemotherapy
Drug: Cisplatin — 75 mg/m² was administered intravenously on Day 1 of each 21-day cycle, infused over a duration of two hours. Treatment with cisplatin was discontinued starting in Cycle 5 and beyond.
Drug: Carboplatin — An area under the curve (AUC) of 5 mg/mL/min was administered intravenously on Day 1 of each 21-day cycle, infused over a duration of 15 to 60 minutes. Treatment with carboplatin was discontinued starting in Cycle 5 and beyond.
Drug: Etoposide — 100 mg/m² was administered intravenously from Day 1 to Day 3 of each 21-day cycle, infused over a duration of 60 minutes. Treatment with etoposide was discontinued starting in Cycle 5 and beyond.
Drug: Placebo — 200 mg was administered intravenously on Day 1 of each 21-day cycle to match tislelizumab.
  Arms: Arm B: Placebo + Chemotherapy

SUMMARY:
This Phase 3 study was a randomized, double-blind, placebo-controlled, multicenter trial designed to evaluate the efficacy of tislelizumab in combination with either cisplatin or carboplatin and etoposide (Arm A), compared to placebo combined with either cisplatin or carboplatin and etoposide (Arm B), as a first-line treatment for participants with previously untreated extensive-stage small cell lung cancer (ES-SCLC).

ELIGIBILITY:
Key Inclusion Criteria:

1. Age≥18 years old, male or female, signed Informed Consent Form (ICF).
2. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
3. Histologically or cytologically confirmed ES-SCLC
4. No prior systemic treatment for ES-SCLC
5. Adequate hematologic and end organ function

Key Exclusion Criteria:

1. Active leptomeningeal disease or uncontrolled, untreated brain metastasis;
2. Prior therapy with an antibody or drug against immune checkpoint pathways, including but not limited to, anti program death receptor-1 (anti-PD-1), anti-PD-L1, or anti cytotoxic T lymphocyte associated antigen 4 (anti CTLA-4) antibody;
3. Was administered a live vaccine ≤ 4 weeks before randomization;
4. Active autoimmune diseases or history of autoimmune diseases that may relapse
5. Any condition that required systemic treatment with either corticosteroids or other immunosuppressive medication ≤ 14 days before randomization;
6. With a history of interstitial lung disease, non-infectious pneumonitis, or uncontrolled systemic diseases;
7. Severe chronic or active infections requiring systemic antibacterial, antifungal or antiviral therapy within 2 weeks prior to randomization, including but not limited to tuberculosis infection;
8. Participant with untreated hepatitis B virus (HBV)/hepatitis C virus (HCV), or a known history of HIV infection;
9. Participants with toxicities (as a result of prior anticancer therapy) which have not recovered to baseline or stabilized at the time of randomization;
10. Clinically significant pericardial effusion, or Clinically uncontrolled pleural effusion

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 457 (Actual)
Dates: Start 2019-07-22 (Actual); Primary Completion 2023-04-19 (Actual); Study Completion 2023-12-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Study Director
Locations (50):
- China (50):
  - The Second Hospital of Anhui Medical University, Hefei, Anhui
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - China Japan Friendship Hospital, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Beijing Hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Chinese Pla General Hospital, Beijing, Beijing Municipality
  - Peking University International Hospital, Beijing, Beijing Municipality
  - Daping Hospital, Third Military Medical University, Chongqing, Chongqing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - The First Hospital of Lanzhou University, Lanzhou, Gansu
  - Cancer Center of Guangzhou Medical University, Guangzhou, Guangdong
  - Guangdong Provincial Peoples Hospital, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Affiliated Hospital of Guilin Medical University, Guilin, Guangxi
  - The Peoples Hospital of Guangxi Zhuang Autonomous Region, Nanning, Guangxi
  - The Tumor Hospital Affiliated to Guangxi Medical University, Nanning, Guangxi
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Wuhan Central Hospital, Wuhan, Hubei
  - Union Hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Tongji Hospital of Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - Changsha Central Hospital, Changsha, Hunan
  - Xiangya Hospital of Central South University, Changsha, Hunan
  - Hunan Cancer Hospital, Changsha, Hunan
  - General Hospital of Eastern Theater Command, Nanjing, Jiangsu
  - Nanjing Chest Hospital, Nanjing, Jiangsu
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Jilin Cancer Hospital, Changchun, Jilin
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - Liaoning Cancer Hospital and Institute, Shenyang, Liaoning
  - Shaanxi Provincial Cancer Hospital, Xi'an, Shaanxi
  - The First Affiliated Hospital of Xian Jiaotong University, Xi'an, Shaanxi
  - Jinan Central Hospital, Jinan, Shandong
  - Shandong Cancer Hospital, Jinan, Shandong
  - The Affiliated Hospital of Qingdao University Branch South, Qingdao, Shandong
  - Yantai Yuhuangding Hospital, Yantai, Shandong
  - Shanghai Chest Hospital, Shanghai, Shanghai Municipality
  - Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality
  - Sichuan Cancer Hospital and Institute, Chengdu, Sichuan
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality
  - Affiliated Cancer Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - Yunnan Cancer Hospital, Kunming, Yunnan
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Cheng Y, Fan Y, Zhao Y, Huang D, Li X, Zhang P, Kang M, Yang N, Zhong D, Wang Z, Yu Y, Zhang Y, Zhao J, Qin T, Chen C, Leaw S, Zheng W, Song Y; RATIONALE-312 Study Group. Tislelizumab Plus Platinum and Etoposide Versus Placebo Plus Platinum and Etoposide as First-Line Treatment for Extensive-Stage SCLC (RATIONALE-312): A Multicenter, Double-Blind, Placebo-Controlled, Randomized, Phase 3 Clinical Trial. J Thorac Oncol. 2024 Jul;19(7):1073-1085. doi: 10.1016/j.jtho.2024.03.008. Epub 2024 Mar 7. PMID 38460751
- [Derived] Cheng Y, Qin T, Chen C, B Barnes F, Barnes G. Tislelizumab plus platinum and etoposide versus placebo plus platinum and etoposide as first-line treatment for extensive-stage small-cell lung cancer: patient-reported outcomes in the RATIONALE-312 trial. Curr Med Res Opin. 2026 Jan 30:1-11. doi: 10.1080/03007995.2026.2620691. Online ahead of print. PMID 41614649
- [Derived] Long R, Chen F. First-line chemotherapy with tislelizumab for patients with extensive-stage small cell lung cancer: a cost-effectiveness analysis. Sci Rep. 2024 Dec 30;14(1):31958. doi: 10.1038/s41598-024-83509-x. PMID 39738721
- [Derived] Wu J, Zhang A, Li L, Liu S, Yang F, Yang R. Meta-analysis of the Efficacy and Tolerability of Immune Checkpoint Inhibitors Combined With Chemotherapy in First-line Treatment of Small Cell Lung Cancer. Clin Ther. 2021 Mar;43(3):582-593.e2. doi: 10.1016/j.clinthera.2020.12.017. Epub 2021 Jan 25. PMID 33509647

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled across multiple study centers in China. The first participant was randomized on July 22, 2019, and the last participant completed the study on December 29, 2023.
Pre-assignment Details: Participants were randomized in a 1:1 ratio to receive chemotherapy (cisplatin or carboplatin + etoposide) in combination with tislelizumab (Arm A) or placebo (Arm B).
Groups:
- Arm A: Tislelizumab + Chemotherapy: Participants received tislelizumab with cisplatin or carboplatin and etoposide every 3 weeks for 4 cycles, then transitioned to maintenance tislelizumab every 3 weeks. Tislelizumab (200 mg) was administered on Day 1 of each cycle. Cisplatin (75 mg/m²) or carboplatin (AUC 5 mg/mL/min) was given on Day 1, and etoposide (100 mg/m²) on Days 1 to 3, with all chemotherapy discontinued after Cycle 4.
- Arm B: Placebo + Chemotherapy: Participants received a placebo (matching the tislelizumab dose) with cisplatin or carboplatin and etoposide every 3 weeks for 4 cycles, then transitioned to maintenance placebo every 3 weeks. Cisplatin (75 mg/m²) or carboplatin (AUC 5 mg/mL/min) was given on Day 1, and etoposide (100 mg/m²) on Days 1 to 3, with all chemotherapy discontinued after Cycle 4.
Period: Overall Study
Arm/Group | Arm A: Tislelizumab + Chemotherapy | Arm B: Placebo + Chemotherapy
Started | 227 | 230
Treated | 227 | 229
Completed (Participants who were still on-study at the time of study completion.) | 49 | 26
Not Completed | 178 | 204
Not completed — Death | 175 | 196
Not completed — Withdrawal by Subject | 1 | 6
Not completed — Lost to Follow-up | 2 | 2

BASELINE CHARACTERISTICS:
Population: The Intent-to-Treat Analysis Set included all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Tislelizumab + Chemotherapy | Arm B: Placebo + Chemotherapy | Total
Number analyzed (Participants) | 227 | 230 | 457
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.5 (7.75) | 60.7 (8.25) | 61.1 (8.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 44 | 85
  Male | 186 | 186 | 372
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 227 | 230 | 457
Eastern Cooperative Oncology Group Performance Status [Count of Participants; unit: Participants] — The ECOG scale assesses disease status from 0 to 5. A score of 0 means fully active with no restrictions, while 1 indicates limitations in strenuous activities but the ability to do light work. Score 2 signifies ambulatory and capable of self-care, yet unable to work, being active for over 50% of waking hours. Score 3 reflects limited self-care, confined to bed or a chair for more than half the day. Score 4 indicates complete disability, with the participant fully bedbound, and score 5 means deceased.
  Participants
    0 | 35 | 34 | 69
    1 | 192 | 196 | 388
Brain Metastases [Count of Participants; unit: Participants]
  Yes | 1 | 4 | 5
  No | 226 | 226 | 452
Chemotherapy [Count of Participants; unit: Participants]
  Cisplatin | 47 | 49 | 96
  Carboplatin | 180 | 181 | 361

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: Defined as the time from the date of randomization to the date of death due to any cause. Median OS was estimated using Kaplan-Meier methodology.
Time Frame: From randomization to the primary completion cut-off on April 19, 2023, the median follow-up was 15.44 months (range: 0.2-44.9) for Arm A and 13.22 months (range: 0.1-40.8) for Arm B.
Population: Intent to treat analysis set
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A: Tislelizumab + Chemotherapy | Arm B: Placebo + Chemotherapy
Number analyzed (Participants) | 227 | 230
Months | 15.5 [13.5 to 17.1] | 13.5 [12.1 to 14.9]
Statistical Analysis 1: Comparison: Arm A: Tislelizumab + Chemotherapy vs Arm B: Placebo + Chemotherapy; The null hypothesis stated that the overall survival in Arm A (Tislelizumab + Chemotherapy) is less than or equal to that in Arm B (the placebo group), while the alternative hypothesis posits that the overall survival in Arm A is greater than that in Arm B; Test type: Superiority; p = 0.0040, Log Rank; Stratified log rank test with ECOG performance status, and investigator chosen platinum as stratification factors; Hazard Ratio (HR) = 0.75, 95% CI 2-sided [0.61 to 0.93] — The hazard ratio was estimated using a stratified Cox regression model with Efron's method for ties, stratified by ECOG performance status and investigator-selected platinum agents, with Arm B as the reference group

2. Secondary Outcome: Progression Free Survival (PFS)
Description: Defined as the time from randomization to the first objectively documented disease progression, or death from any cause, whichever occurred first, as assessed by the investigator per the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. Kaplan-Meier methodology was used to estimate the median PFS.
  Progressive Disease (PD): At least a 20% increase in the size of target lesions, with an absolute increase of at least 5 mm, or unequivocal progression of existing non-target lesions, or any new lesions.
Time Frame: as for outcome 1
Population: Intent to treat analysis set
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A: Tislelizumab + Chemotherapy | Arm B: Placebo + Chemotherapy
Number analyzed (Participants) | 227 | 230
Months | 4.7 [4.3 to 5.5] | 4.3 [4.2 to 4.4]
Statistical Analysis 1: Comparison: Arm A: Tislelizumab + Chemotherapy vs Arm B: Placebo + Chemotherapy; Test type: Superiority; p < 0.0001, Log Rank; One-sided log-rank test p-value, stratified by ECOG performance status (1 vs 0) and type of platinum therapy (carboplatin vs cisplatin); Hazard Ratio (HR) = 0.64, 95% CI 2-sided [0.52 to 0.78] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Overall Response Rate (ORR)
Description: Orr is defined as the percentage of participants who had partial response or complete response as determined by the investigator per RECIST v1.1 in all randomized patients with measurable disease at baseline.
  Complete Response (CR): Disappearance of all target and non-target lesions and no new lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm.
  Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions with no progression of non-target lesions and no new lesions, or disappearance of all target lesions with persistence of one or more non-target lesion(s) and/or maintenance of tumor marker level above the normal limits and no new lesions.
Time Frame: as for outcome 1
Population: Intent to treat analysis set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A: Tislelizumab + Chemotherapy | Arm B: Placebo + Chemotherapy
Number analyzed (Participants) | 227 | 230
percentage of participants | 68.3 [61.8 to 74.3] | 61.7 [55.1 to 68.0]
Statistical Analysis 1: Comparison: Arm A: Tislelizumab + Chemotherapy vs Arm B: Placebo + Chemotherapy; Test type: Other; Odds Ratio (OR) = 1.33, 95% CI 2-sided [0.90 to 1.96] — Odds ratio was calculated using Cochran-Mantel-Haenszel estimates and stratified by ECOG performance (1 vs 0) and platinum (Carboplatin vs Cisplatin)

4. Secondary Outcome: Disease Control Rate (DCR)
Description: Defined as the percentage of participants whose best overall response (BOR) is complete response, partial response, or stable disease per RECIST v1.1.
  Stable Disease: Neither sufficient shrinkage of target lesions to qualify for PR nor sufficient increase to qualify for progressive disease, persistence of one or more non-target lesion(s) and/or maintenance of tumor marker level above the normal limits, and no new lesions.
Time Frame: as for outcome 1
Population: Intent to treat analysis set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A: Tislelizumab + Chemotherapy | Arm B: Placebo + Chemotherapy
Number analyzed (Participants) | 227 | 230
percentage of participants | 88.5 [83.7 to 92.4] | 88.3 [83.4 to 92.1]

5. Secondary Outcome: Clinical Benefit Rate (CBR)
Description: Defined as the percentage of participants whose best overall response (BOR) is complete response, partial response, or durable stable disease (stable disease for at least 24 weeks) per RECIST v1.1.
Time Frame: as for outcome 1
Population: Intent to treat analysis set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A: Tislelizumab + Chemotherapy | Arm B: Placebo + Chemotherapy
Number analyzed (Participants) | 227 | 230
percentage of participants | 69.2 [62.7 to 75.1] | 65.2 [58.7 to 71.4]

6. Secondary Outcome: Duration of Response (DOR)
Description: Defined as the time from the first occurrence of a documented objective response to the time of relapse, as determined by the investigator per RECIST v1.1, or death from any cause, whichever comes first. Median DOR was estimated using Kaplan-Meier methodology.
Time Frame: as for outcome 1
Population: Intent to treat analysis Set. Only participants with best overall response of complete response or partial response confirmed per RECIST v1.1 were included in the analysis, and percentages were based on the number of responders
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A: Tislelizumab + Chemotherapy | Arm B: Placebo + Chemotherapy
Number analyzed (Participants) | 155 | 142
Months | 4.3 [4.1 to 5.6] | 3.7 [3.0 to 4.1]

7. Secondary Outcome: Number of Participants With Adverse Events
Description: Number of participants with treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs) graded according to the National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0.
Time Frame: From the first dose to 30 days after the last dose or final cutoff on December 29, 2023, maximum treatment exposure was 232 weeks for Arm A and 157 weeks for Arm B.
Population: The Safety Analysis Set includes all participants randomized and received any dose of any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Tislelizumab + Chemotherapy | Arm B: Placebo + Chemotherapy
Number analyzed (Participants) | 227 | 229
Participants
  TEAEs | 226 | 228
  SAEs | 94 | 70

8. Secondary Outcome: Change From Baseline in the European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) Global Health Status and Physical Function Score.
Description: The EORTC QLQ-30 contains 30 questions that incorporate 5 functional scales (physical functioning, role functioning, emotional functioning, cognitive functioning, and social functioning), 1 global health status scale, 3 symptom scales (fatigue, nausea and vomiting, and pain), and 6 single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). The participant answers questions about their health during the past week. There are 28 questions answered on a 4-point scale where 1 = Not at all (best) and 4 = Very Much (worst) and 2 global health quality of life (QOL) questions answered on a 7-point scale where 1 = Very poor and 7 = Excellent. Raw scores are transformed into a 0 to 100 scale via linear transformation. Higher scores in GHS and functional scales indicate better quality of life.
Time Frame: Baseline to Cycles 4 and 6 ( Each cycle was 21 days)
Population: The HRQoL analysis set included all randomized participants who received any dose of study drug and completed at least one HRQoL assessment. Only participants with data at both baseline and corresponding post-baseline visit are included in the analysis at each time point.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Arm A: Tislelizumab + Chemotherapy | Arm B: Placebo + Chemotherapy
Number analyzed (Participants) | 225 | 229
Score on a scale
  Global Health Status/Quality of Life (Cycle 4): number analyzed (Participants) | 190 | 202
  Global Health Status/Quality of Life (Cycle 4) | 8.9 (22.79) | 4.5 (19.46)
  Global Health Status/Quality of Life (Cycle 6): number analyzed (Participants) | 152 | 160
  Global Health Status/Quality of Life (Cycle 6) | 11.3 (21.30) | 4.2 (19.04)
  Physical Functioning (Cycle 4): number analyzed (Participants) | 190 | 202
  Physical Functioning (Cycle 4) | 0.6 (14.82) | 0.4 (14.57)
  Physical Functioning (Cycle 6): number analyzed (Participants) | 152 | 160
  Physical Functioning (Cycle 6) | 1.9 (15.18) | 1.8 (12.36)

9. Secondary Outcome: Change From Baseline in European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire-Lung Cancer (EORTC QLQ-LC13) Symptom Scores
Description: Change from baseline in EORTC QLQ-CL13 scores for coughing, dysphagia, and chest pain. The EORTC QLQ-LC13 is a questionnaire that measures lung cancer-specific disease and treatment symptoms. It includes questions about specific symptoms in which participants respond based on a 4-point scale, where 1 is "not at all" and 4 is "very much". Raw scores are transformed into a 0 to 100 scale via linear transformation. A lower score indicates an improvement in symptoms.
Time Frame: Baseline to Cycles 4 and 6 ( Each cycle was 21 days)
Population: HRQoL analysis set. Only participants with data at both baseline and corresponding post-baseline visit are included in the analysis at each time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm A: Tislelizumab + Chemotherapy | Arm B: Placebo + Chemotherapy
Number analyzed (Participants) | 225 | 229
score on a scale
  Coughing (Cycle 4): number analyzed (Participants) | 190 | 202
  Coughing (Cycle 4) | -19.5 (26.58) | -16.0 (22.85)
  Coughing (Cycle 6): number analyzed (Participants) | 152 | 160
  Coughing (Cycle 6) | -18.6 (27.86) | -16.7 (25.08)
  Dysphagia (Cycle 4): number analyzed (Participants) | 190 | 202
  Dysphagia (Cycle 4) | -2.5 (12.12) | -3.1 (14.72)
  Dysphagia (Cycle 6): number analyzed (Participants) | 152 | 160
  Dysphagia (Cycle 6) | -2.9 (11.47) | -3.5 (15.23)
  Chest Pain (Cycle 4): number analyzed (Participants) | 190 | 202
  Chest Pain (Cycle 4) | -7.5 (22.65) | -5.9 (20.97)
  Chest Pain (Cycle 6): number analyzed (Participants) | 152 | 160
  Chest Pain (Cycle 6) | -7.0 (25.34) | -6.9 (21.51)

10. Secondary Outcome: Time to Deterioration (TTD)
Description: Time to deterioration is defined as the time from randomization to the first confirmed worsening score or death. Clinically meaningful deterioration is defined as a ≥10-point decrease from baseline in QLQ-C30 physical functioning and a ≥10-point increase in QLQ-LC13 coughing and chest pain scores. If a participant did not have an event (death or deterioration), they were censored at their last clinic visit at which corresponding score was measured. Median TTD was estimated using Kaplan-Meier methodology.
Time Frame: From randomization to the primary completion data cut-off on April 19, 2023, the median follow-up was 15.44 months (range: 0.2-44.9) for Arm A and 13.22 months (range: 0.1-40.8) for Arm B.
Population: HRQoL analysis set
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A: Tislelizumab + Chemotherapy | Arm B: Placebo + Chemotherapy
Number analyzed (Participants) | 227 | 229
Months
  QLQ-C30: Physical Functioning | NA [20.5 to NA] — Could not be estimated due to insufficient number of participants with events | NA [10.3 to NA] — Could not be estimated due to insufficient number of participants with events
  QLQ-LC13: Coughing | NA [NA to NA] — Could not be estimated due to insufficient number of participants with events | NA [NA to NA] — Could not be estimated due to insufficient number of participants with events
  QLQ-LC13: Chest Pain | NA [NA to NA] — Could not be estimated due to insufficient number of participants with events | NA [NA to NA] — Could not be estimated due to insufficient number of participants with events
Statistical Analysis 1: Comparison: Arm A: Tislelizumab + Chemotherapy vs Arm B: Placebo + Chemotherapy; Analyses of Time to Deterioration of EORTC QLQ-C30 Physical Functioning Score; Test type: Other; Hazard Ratio (HR) = 0.92, 95% CI 2-sided [0.642 to 1.330] — Hazard ratio was based on unstratified Cox regression model including treatment as covariate
Statistical Analysis 2: Comparison: Arm A: Tislelizumab + Chemotherapy vs Arm B: Placebo + Chemotherapy; Analyses of Time to Deterioration of EORTC QLQ-LC13 Coughing Score; Test type: Other; Hazard Ratio (HR) = 0.73, 95% CI 2-sided [0.473 to 1.123] — Hazard ratio was based on unstratified Cox regression model including treatment as covariate
Statistical Analysis 3: Comparison: Arm A: Tislelizumab + Chemotherapy vs Arm B: Placebo + Chemotherapy; Analyses of Time to Deterioration of EORTC QLQ-LC13 Chest Pain Score; Test type: Other; Hazard Ratio (HR) = 0.72, 95% CI 2-sided [0.485 to 1.057] — Hazard ratio was based on unstratified Cox regression model including treatment as covariate

ADVERSE EVENTS:
Time Frame: All-cause mortality is reported from randomization to the end of study (up to 53 months). Adverse events are reported from from the first dose to 30 days after the last dose or final cutoff on December 29, 2023, maximum treatment exposure was 232 weeks for Arm A and 157 weeks for Arm B.
Description: All-cause mortality is reported for all randomized participants. Serious and other adverse events includes all randomized participants who received ≥ 1 dose of any study treatment.
Arm/Group | Arm A: Tislelizumab + Chemotherapy | Arm B: Placebo + Chemotherapy
All-Cause Mortality (participants affected / at risk) | 175/227 | 196/230
Serious Adverse Events (participants affected / at risk) | 94/227 | 70/229
Other Adverse Events (participants affected / at risk) | 226/227 | 228/229
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Tislelizumab + Chemotherapy (N=227) | Arm B: Placebo + Chemotherapy (N=229)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 4 (4)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (3) | 5 (5)
Leukopenia (Blood and lymphatic system disorders) | 3 (3) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 16 (18) | 9 (9)
Thrombocytopenia (Blood and lymphatic system disorders) | 17 (20) | 18 (20)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Autoimmune myocarditis (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1)
Immune-mediated myocarditis (Cardiac disorders) | 3 (3) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Deafness neurosensory (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 2 (2) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 3 (3) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 2 (2) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0)
Subileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0)
Death (General disorders) | 2 (2) | 0 (0)
Disease progression (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 2 (2) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 0 (0)
Immune-mediated hepatitis (Hepatobiliary disorders) | 2 (2) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Encephalitis (Infections and infestations) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Infectious pleural effusion (Infections and infestations) | 1 (1) | 0 (0)
Phlebitis infective (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 4 (4) | 5 (5)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Upper respiratory tract infection bacterial (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 4 (4) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 3 (3) | 0 (0)
Neutrophil count decreased (Investigations) | 5 (6) | 3 (3)
Platelet count decreased (Investigations) | 5 (6) | 5 (6)
Troponin T increased (Investigations) | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 5 (5) | 3 (3)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Diabetic ketosis (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 5 (6) | 1 (1)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Paraneoplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Brain oedema (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 2 (2) | 0 (0)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0)
Intracranial pressure increased (Nervous system disorders) | 0 (0) | 1 (1)
Meningitis noninfective (Nervous system disorders) | 1 (1) | 0 (0)
Neuritis (Nervous system disorders) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 2 (2) | 0 (0)
Secondary cerebellar degeneration (Nervous system disorders) | 1 (1) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (5)
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Immune-mediated dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Circulatory collapse (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Superior vena cava syndrome (Vascular disorders) | 0 (0) | 1 (1)
Vena cava thrombosis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Tislelizumab + Chemotherapy (N=227) | Arm B: Placebo + Chemotherapy (N=229)
Anaemia (Blood and lymphatic system disorders) | 192 (356) | 191 (329)
Leukopenia (Blood and lymphatic system disorders) | 74 (205) | 55 (173)
Neutropenia (Blood and lymphatic system disorders) | 149 (445) | 157 (492)
Thrombocytopenia (Blood and lymphatic system disorders) | 108 (247) | 114 (248)
Sinus tachycardia (Cardiac disorders) | 10 (13) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 17 (21) | 1 (1)
Hypothyroidism (Endocrine disorders) | 28 (38) | 9 (10)
Abdominal distension (Gastrointestinal disorders) | 14 (15) | 8 (10)
Abdominal pain (Gastrointestinal disorders) | 7 (8) | 5 (5)
Abdominal pain upper (Gastrointestinal disorders) | 16 (20) | 7 (8)
Constipation (Gastrointestinal disorders) | 84 (136) | 58 (84)
Diarrhoea (Gastrointestinal disorders) | 36 (49) | 31 (38)
Dysphagia (Gastrointestinal disorders) | 5 (5) | 7 (10)
Gingival pain (Gastrointestinal disorders) | 10 (10) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 7 (8) | 0 (0)
Nausea (Gastrointestinal disorders) | 101 (193) | 100 (171)
Oral pain (Gastrointestinal disorders) | 2 (2) | 8 (14)
Toothache (Gastrointestinal disorders) | 11 (16) | 7 (7)
Vomiting (Gastrointestinal disorders) | 56 (93) | 54 (85)
Asthenia (General disorders) | 17 (20) | 16 (19)
Chest discomfort (General disorders) | 14 (19) | 6 (6)
Face oedema (General disorders) | 9 (9) | 3 (3)
Fatigue (General disorders) | 27 (33) | 14 (15)
Malaise (General disorders) | 29 (42) | 31 (40)
Non-cardiac chest pain (General disorders) | 18 (22) | 17 (18)
Oedema peripheral (General disorders) | 11 (12) | 11 (13)
Pyrexia (General disorders) | 30 (35) | 17 (22)
Pneumonia (Infections and infestations) | 5 (6) | 13 (13)
Upper respiratory tract infection (Infections and infestations) | 17 (25) | 9 (9)
Infusion related reaction (Injury, poisoning and procedural complications) | 8 (10) | 5 (5)
Alanine aminotransferase increased (Investigations) | 67 (129) | 46 (62)
Aspartate aminotransferase increased (Investigations) | 51 (85) | 35 (60)
Bilirubin conjugated increased (Investigations) | 7 (10) | 4 (4)
Blood alkaline phosphatase increased (Investigations) | 13 (19) | 11 (14)
Blood bilirubin increased (Investigations) | 16 (32) | 7 (11)
Blood creatine phosphokinase MB increased (Investigations) | 11 (15) | 9 (11)
Blood creatine phosphokinase increased (Investigations) | 26 (48) | 6 (12)
Blood creatinine increased (Investigations) | 19 (31) | 14 (26)
Blood lactate dehydrogenase increased (Investigations) | 14 (16) | 12 (18)
Fibrin D dimer increased (Investigations) | 5 (6) | 7 (7)
Gamma-glutamyltransferase increased (Investigations) | 27 (45) | 21 (30)
Lymphocyte count decreased (Investigations) | 25 (68) | 28 (62)
Neutrophil count decreased (Investigations) | 50 (151) | 56 (220)
Platelet count decreased (Investigations) | 31 (52) | 35 (80)
Weight decreased (Investigations) | 24 (26) | 12 (12)
Weight increased (Investigations) | 19 (27) | 8 (8)
White blood cell count decreased (Investigations) | 126 (388) | 147 (478)
Decreased appetite (Metabolism and nutrition disorders) | 88 (149) | 86 (141)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 11 (21) | 14 (23)
Hyperglycaemia (Metabolism and nutrition disorders) | 28 (65) | 22 (35)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 22 (51) | 19 (29)
Hyperuricaemia (Metabolism and nutrition disorders) | 31 (61) | 22 (32)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 54 (83) | 44 (69)
Hypocalcaemia (Metabolism and nutrition disorders) | 19 (25) | 12 (13)
Hypochloraemia (Metabolism and nutrition disorders) | 20 (27) | 13 (14)
Hypokalaemia (Metabolism and nutrition disorders) | 39 (82) | 19 (26)
Hypomagnesaemia (Metabolism and nutrition disorders) | 11 (25) | 4 (4)
Hyponatraemia (Metabolism and nutrition disorders) | 55 (88) | 56 (83)
Hypophosphataemia (Metabolism and nutrition disorders) | 9 (27) | 8 (11)
Arthralgia (Musculoskeletal and connective tissue disorders) | 34 (44) | 18 (23)
Back pain (Musculoskeletal and connective tissue disorders) | 17 (20) | 22 (25)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 26 (35) | 18 (27)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 (13) | 14 (20)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 (17) | 12 (17)
Dizziness (Nervous system disorders) | 24 (33) | 19 (21)
Headache (Nervous system disorders) | 23 (27) | 11 (12)
Hypoaesthesia (Nervous system disorders) | 10 (13) | 4 (4)
Insomnia (Psychiatric disorders) | 39 (58) | 26 (33)
Cough (Respiratory, thoracic and mediastinal disorders) | 37 (41) | 27 (33)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 24 (27) | 27 (27)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 23 (31) | 25 (32)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 11 (11) | 9 (17)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 5 (5)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 22 (24) | 11 (13)
Alopecia (Skin and subcutaneous tissue disorders) | 180 (182) | 182 (185)
Pruritus (Skin and subcutaneous tissue disorders) | 15 (18) | 6 (8)
Rash (Skin and subcutaneous tissue disorders) | 33 (44) | 20 (24)
Hypertension (Vascular disorders) | 21 (51) | 18 (28)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
BeiGene has 18 months from the end of the study at all sites to publish overall study results. After the 1st multi-site publication or the expiration of publication period, Investigators are free to publish/present the results of the study. Investigators must submit all draft publications/presentations to us for review 60 days prior to the planned publication/presentation date. BeiGene may request deletion of its confidential information & may request a further delay to protect its IP rights.

DOCUMENTS (2):
  • Study Protocol (2020-09-02): https://cdn.clinicaltrials.gov/large-docs/16/NCT04005716/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-24): https://cdn.clinicaltrials.gov/large-docs/16/NCT04005716/SAP_001.pdf